CLINICAL TRIAL: NCT06546371
Title: Spinal Cord Stimulation for Intractable Mononeuropathy: a Pilot Study
Brief Title: Spinal Cord Stimulation for Intractable Mononeuropathy
Acronym: SCIMONO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Frank Huygen, Head of Centre for Pain Medicine, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2023-0644
Record Dates: First submitted 2024-06-22; First posted 2024-08-09 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Mononeuropathies; Spinal Cord Stimulation
MeSH Terms: conditions — Mononeuropathies

STUDY DESIGN:
Intervention Model Description: Mono-center explorative pilot study in 12 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Spinal cord stimulation (Experimental): Patients are all included in this experimental arm, where they receive all four stimulation options consecutively, but in different orders. After receiving all four stimulation options, the patients are allowed to choose which stimulation option of the four they want to have for the following period.
  Interventions: Device: Spinal cord stimulator

INTERVENTIONS:
Device: Spinal cord stimulator — Electrical stimulation of the dorsal horn to reduce chronic pain.

SUMMARY:
Rationale: For patients with mononeuropathy, literature has shown that spinal cord stimulation (SCS) is an effective therapy for patients who are therapy-resistant to more conventional treatments. However, there is a strong need for higher quality evidence to determine the place of this therapy in this target group. Before conducting a large randomized controlled trial (RCT) we propose to conduct an explorative pilot study based on which an effect size estimation and power calculation for a larger study can be done. We will assess the effects of SCS in patients with mononeuropathy measured according to the "Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials" (IMMPACT) guidelines, and assess the stimulation paradigm preferences in these patients.

Objective: To perform an explorative pilot study based on which an effect size estimation and power calculation for an efficacy trial can be done.

Study design: Mono-center explorative pilot study in 12 patients with intractable peripheral mononeuropathic pain who receive a spinal cord stimulator at the Erasmus Medical Centre.

Study population: 12 patients suffering from intractable peripheral mononeuropathic pain.

Intervention: Participants who receive a spinal cord stimulator must fill in IMMPACT guideline questionnaires and undergo several measurement procedures after receiving SCS implantation. The effect of various SCS paradigms on the chronic mononeuropathic pain is assessed at 3 and 6 months.

Main study parameters/endpoints: Effect of 6 months of individually optimized SCS in patients with mononeuropathy according to the IMMPACT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from painful intractable peripheral mononeuropathy in the distal extremities, preferably post-traumatic or post-surgical, confirmed by electromyography (EMG)
* Symptoms refractory to conventional medical management for at least 6 months according to treating physician
* 18 years or older
* Pain score on numeric rating scale (NRS) of at least 5 (average pain intensity in week prior to assessment)
* Stable or absent concomitant analgesics

Exclusion Criteria:

* Mononeuropathy located in the head or torso
* Mononeuropathy by avulsion at the plexus brachialis
* Life expectancy <1 year
* Anticoagulant drug therapy or disturbed coagulation
* Immune-compromised patients
* Pregnancy
* Lack of cooperation of the patient or patient has a history of noncompliance with regard to (a) medical regime(s)
* Patients with psychological factors or addiction that require treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Effect of spinal cord stimulation (SCS) in patients with mononeuropathy as assessed by the perceived pain intensity. | 6 months
  Perceived pain intensity as assessed by the brief pain inventory (BPI), with pain scores where 0 is no pain and 10 is worst pain imaginable.

SECONDARY OUTCOMES:
Effect of SCS in patients with mononeuropathy as assessed by quantitative sensory testing (QST). | 6 months
  Quantitative sensory testing (QST) measures sensory thresholds for pain, touch, vibration, and temperature sensations, with the main goal to assess sensory functioning.
Effect of SCS in patients with mononeuropathy on quality of life. | 6 months
  Quality of life as assessed by the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire.
Patient preferences for SCS paradigms as assessed by the perceived pain intensity. | 3 months
  Perceived pain intensity as assessed by the brief pain inventory (BPI), with pain scores where 0 is no pain and 10 is worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Centre, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes